CLINICAL TRIAL: NCT06407986
Title: Pulmonary Ventilation Heterogeneity Determined by Electrical Impedance Tomography During Pulmonary Function Testing in Subjects With Normal One-second Rates
Brief Title: Pulmonary Ventilation Heterogeneity Determined by EIT During PFT in Subjects With Normal One-second Rates
Status: Recruiting | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: '2023-933-01'
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Lung Function Decreased
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal lung function: After using a bronchodilator, FEV1/FVC ≥70%, FEV1 and FVC ≥80% of reference values.
  Interventions: Diagnostic Test: pulmonary function test
- Preserved ratio impaired spirometry: After using a bronchodilator, FEV1/FVC≥70%, FEV1 and/or FVC<80% of reference values.
  Interventions: Diagnostic Test: pulmonary function test

INTERVENTIONS:
Diagnostic Test: pulmonary function test — Whether the estimated value of FEV1 and FVC is greater than 80%.

SUMMARY:
To evaluate the demographic characteristics of normal one-second rates population in patients with pulmonary function tests recommended by outpatient physicians.

To investigate whether EIT can identify spatial and temporal heterogeneity of lung ventilation in individuals with normal one-second rates during pulmonary function testing.

To investigate the distribution patterns of lung ventilation in individuals with normal one-second rates using this technique, and provide references and evidence for early screening, diagnosis, treatment monitoring, and prognostic evaluation.

DETAILED DESCRIPTION:
In the GOLD 2023 guidelines, a newly introduced term called "Preserved Ratio Impaired Spirometry (PRISm)" refers to patients who have a normal forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) ratio (FEV1/FVC≥0.7, after bronchodilator use), but exhibit impaired pulmonary ventilation function with FEV1 and/or FVC values below 80% of the predicted value. In the past, these patients were often classified as GOLD U or restrictive ventilatory impairment. In recent years, several large cross-sectional and longitudinal studies on PRISm have revealed its high prevalence, ranging from 5-20% due to population heterogeneity. Notably, approximately 10% to 40% of patients with PRISm tend to develop chronic obstructive pulmonary disease (COPD), resulting in frequent healthcare utilization. Moreover, subjects with normal lung function are also at risk of converting to PRISm during long-term follow-up. Studies have found that such patients are associated with increased respiratory symptoms, reduced quality of life, and increased burden of cardiovascular disease. A recent meta-analysis showed a significant increased risk of all-cause, cardiovascular, and respiratory-related mortality risk in PRISm patients. Currently, there are no diagnostic and treatment guidelines for PRISm, but studies highlights the importance of screening and identifying PRISm, with follow-up and early intervention if necessary.

Electrical Impedance Tomography (EIT) is an emerging imaging technology developing rapidly in recent years, with many advantages such as non-invasive, non-radiation and simple operation. Its principle is to measure the voltage or current signals through electrodes on the body surface, and then reconstructing images of the distribution of impedance changes. This technology is widely used in pulmonary diseases, including monitoring lung ventilation distribution, blood perfusion, and titration of positive end-expiratory pressure. EIT images have high spatial and temporal resolution, can display physiological and pathological changes in real time based on breathing. In 2022, China issued the clinical application consensus of electrical impedance tomography in critical respiratory management, further promoting the application of this technology in respiratory management. However, the number of clinical studies on EIT in identifying airway obstruction in COPD patients is limited. It has been proven that in COPD patients, EIT combined with pulmonary function tests can evaluate the spatial and temporal distribution of lung capacity in different regions and identify pathologically induced ventilation heterogeneity. At present, the pathophysiological mechanism of PRISm is still under discussion. Studies have found that PRISm is related to small airway dysfunction (SAD) and decreased total lung capacity. Computed Tomography (CT) can be used to evaluate small airway function and observe the morphological and structural changes of lung tissue, but it has but it has some disadvantages such as long duration and radiation exposure. Therefore, EIT may be a good choice for rapidly assessing regional lung function in PRISm patients. Due to the scarcity of EIT in PRISm studies, investigators have initiated a clinical study to evaluate whether ventilation heterogeneity in PRISm patients can be obtained through the combination of EIT and pulmonary function tests.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years old. Patients who need to complete lung function tests assessed by outpatient physicians.

Patients willing to participate in the study and sign an informed consent form.

Exclusion Criteria:

Patients with FEV1/FVC less than 0.7 after a bronchiectasis test. Patients with a history of lung diseases other than COPD, previous lung surgery, or radiation therapy.

Patients who cannot be evaluated for EIT or who interfere with EIT results, such as implanted pacemakers/cardioverters.

Patients who cannot complete EIT or may interfere with EIT results, such as those with implanted pacemakers/defibrillators.

Patients who cannot complete lung function tests, such as myocardial infarction or shock in the past 3 months; severe heart failure or angina in the past 4 weeks，uncontrolled hypertension (systolic >200mmHg, diastolic >100mmHg)，severe hyperthyroidism etc.

Vulnerable populations, including patients with mental illnesses, cognitive impairments, critically ill patients, illiterate, pregnant women, etc.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After using a bronchodilator, FEV1/FVC ≥70%.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
regional FEV1 | one month
  They were calculated for each pixel within the lung areas by EIT data analysis
regional FVC | one month
  They were calculated for each pixel within the lung areas by EIT data analysis

SECONDARY OUTCOMES:
St. George's Respiratory Questionnaire | one month
  Score change，the higher the score, the more severe the symptoms
regional obstructive ratio（rOR） | one month
  It was calculated based on the size of obstructed regions in related to the entire lung area.

CONTACTS AND LOCATIONS:
Overall Officials: Huiqing Ge, Study Chair — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No